CLINICAL TRIAL: NCT04578041
Title: An Open Label Pilot Study to Investigate the Effect of Transcranial Rotating Permanent Magnetic Stimulation (TRPMS) on Gait, Balance and Depression in People With Multiple Sclerosis (MS)
Brief Title: TRPMS to Improve Mobility and Depression in Multiple Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01101
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
Keywords: Transcranial Rotating Permanent Magnetic Stimulation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1: TRPMS + Aerobic Physical Activity Program (Experimental)
  Interventions: Device: TRPMS (Transcranial Rotating Permanent Magnet Stimulation); Other: Aerobic Exercise Program
- Arm 2: TRPMS + Adaptive Cognitive Training (Active Comparator)
  Interventions: Device: TRPMS (Transcranial Rotating Permanent Magnet Stimulation); Other: Computerized CT (Cognitive Training)

INTERVENTIONS:
Device: TRPMS (Transcranial Rotating Permanent Magnet Stimulation) — TRPMS ( is administered through a head cap worn by the participant and controlled by QHTimeStimulate application via computer tablet.
  * Modality: Excitatory stimulation
  * Frequency: 5 Hz
  * Interval between stimulus: 100 ms
  * Duration of each stimulus: 25 ms
  * Duration of stimulation: 40 minutes
  * Position of microstimulators: over primary motor cortex and supplementary motor area for Arm 1; over left and right dorsolateral prefrontal cortex for Arm 2
Other: Aerobic Exercise Program — Aerobic exercise consisting of 40 minutes of cycling training with a seated elliptical machine. The daily physical activity program will consist of three 10-minute bouts of aerobic exercise interspersed with two 5-minute bouts of rest. The participants will exercise maintaining their Heart Rate (HR) at least between 60-80% of the maximum age-related HR.
  Arms: Arm 1: TRPMS + Aerobic Physical Activity Program
Other: Computerized CT (Cognitive Training) — Computerized cognitive training (CT) consisting of 40 minutes Brain-HQ training.
  The adaptive cognitive training games also serve to engage them during the stimulation session, and to keep them seated at the computer for the entire duration of the session.
  Arms: Arm 2: TRPMS + Adaptive Cognitive Training

SUMMARY:
This study is aimed to test the efficacy of 10 sessions of Transcranial Rotating Permanent Magnetic Stimulation (TRPMS) paired with aerobic exercise or computerized cognitive training (CT) on mobility and depression symptoms in 40 individuals affected by multiple sclerosis (MS).

Participants in Arm 1 will complete 10x40 minutes daily sessions of TRPMS+aerobic exercise. Participants in Arm 2 will complete TRPMS+computerized CT. Primary outcomes for both arms will be assessed at baseline, at treatment end and after 4-week from the treatment end (follow-up).

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in Arm 1 of this study, an individual must meet all of the following criteria:

1. Between ages 18 - 70
2. SDMT z-score ≥ -3.0
3. Wide Range Achievement Test-4th Edition (WRAT-4) Reading Recognition scaled score ≥ 85
4. Definite MS diagnosis as assessed by a licensed physician (all subtypes - RRMS, PPMS, SPMS)
5. Expanded Disability Status Scale (EDSS) ≤ 6.5
6. Clinically stable disease course with absence of relapse within the past 30 days
7. Able to understand the informed consent process and provide consent to participate in the study
8. Complete the TMS screening questionnaire
9. Able to commit to study timeframe
10. Clinically significant gate deviations (T25-FW > 5.0 seconds)
11. Able to walk independently with or without assistive device (i.e. cane, crutches, or walking frames) for medium distance
12. Able to exercise with seated elliptical machine

In order to be eligible to participate in Arm 2 of this study, an individual must meet all of the following criteria:

1. Between ages 18 - 70
2. SDMT z-score ≥ -3.0
3. Wide Range Achievement Test-4th Edition (WRAT-4) Reading Recognition scaled score ≥ 85
4. Definite MS diagnosis as assessed by a licensed physician (all subtypes - RRMS, PPMS, SPMS)
5. Expanded Disability Status Scale (EDSS) ≤ 6.5
6. Clinically stable disease course with absence of relapse within the past 30 days
7. Able to understand the informed consent process and provide consent to participate in the study
8. Complete the TMS screening questionnaire
9. Able to commit to study timeframe
10. Elevated symptoms of depression as determined by BDI of ≥ 4

Exclusion Criteria:

1. Visual, auditory or motor deficits that would influence participant safety as assessed by a licensed physician
2. History of seizure or epileptic history as assessed by licensed physician
3. Medication which significantly lower the seizure threshold as assessed by licensed physician
4. Primary psychiatric disorder that would influence ability to participate
5. Uncontrolled headaches and migraine or recent changes in the rate or severity of head pressure, headache, or migraine in the past two weeks
6. History of stroke or head trauma (e.g., head injury, brain surgery) or medical device implanted in the head (e.g. Deep Brain Stimulator) or in the neck (e.g. Vagus Nerve Stimulator)
7. History of uncontrolled or labile hypertension
8. Other serious uncontrolled medical condition or recent medical traumas
9. Presence of metal or electronic implants in the body contraindicated for TMS
10. Alcohol or other substance use disorder
11. Pregnant or breastfeeding
12. History of clinically significant abnormalities on electrocardiogram (EKG) (Arm 1 only)
13. Presence of chronic medical illness and/or severe ataxia (Arm 1 only)
14. Functional surgery for lower limb in the past 6 months (e.g. hip or knee replacement) (Arm 1 only)
15. Lower limb Botulinum toxin injection within the past 2 months (Arm 1 only)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Percent of Sessions Completed | Day 10
  Feasibility of at-home usage of TRPMS device measured by percent of sessions completed (80%)
Change in Gait Velocity | Baseline (Day 0), Day 10
  To determine the primary efficacy of the TRPMS intervention paired with aerobic exercise, gait velocity will be assessed during the instrumented 10-meter walking test. Gait velocity will be measured using a wearable inertial sensor (G-Sensor).
Change in PROMIS Depression Score | Baseline (Day 0), Day 10
  Arm 2: To determine the primary efficacy of the TRPMS intervention paired with computerized CT, changes in PROMIS Depression from baseline to treatment-end will be measured. The PROMIS Depression questionnaire consists of 8 items. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.

SECONDARY OUTCOMES:
Change in Gait Velocity | Baseline (Day 0), Week 4
  Arm 1: To assess sustained improvements, gait velocity will be assessed during the instrumented 10-meter walking test. Gait velocity will be measured using a wearable inertial sensor (G-Sensor).
Change in Distance Traveled During 2-Minute Walking Test | Baseline (Day 0), Day 10
  Arm 1
Change in the Total Time for Completing the Timed Up and Go (TUG) test | Baseline (Day 0), Day 10
  Arm 1: The test requires the subject to rise from a chair, walk 3.0 m at a comfortable pace to a mark placed on the floor, turn around at the 3.0 m mark, walk back to the starting point, and return to sitting in the chair.
Change in Modified Fatigue Impact Scale (MFIS) Score | Baseline (Day 0), Day 10
  MFIS consists of 21 statements that describe the effects of fatigue. Each statement is scored on a scale of 0-4 (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = almost always). The total MFIS score can range from 0-84; the higher the score, the stronger the feelings of fatigue.
Change in Short Form (SF)-36 Score | Baseline (Day 0), Day 10
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Change in PROMIS Depression Score | Baseline (Day 0), Week 4
  Arm 2: To determine the primary efficacy of the TRPMS intervention paired with computerized CT, changes in PROMIS Depression from baseline to treatment-end will be measured. The PROMIS Depression questionnaire consists of 8 items. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Change in Center for Epidemiological Studies-Depression short form (CESD-10) Score | Baseline (Day 0), Day 10
  Arm 2: CESD-10 10-item Likert scale questionnaire assessing depressive symptoms in the past week. It includes three items on depressed affect, five items on somatic symptoms, and two on positive affect. Options for each item range from "rarely or none of the time" (score of 0) to "all of the time" (score of 3). The total range of score is 0-30; higher scores indicate the presence of significant depressive symptoms.
Change in Patient Health Questionnaire 9 (PHQ-9) Score | Baseline (Day 0), Day 10
  Arm 2: The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). A PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
Change in Inventory of Depressive Symptomatology Self-Report (IDS-SR) Score | Baseline (Day 0), Day 10
  Arm 2: Each of the 28 items is scored on a 1 to 3 scale (0-the absence of pathology; 3-severe pathology). The total scores range from 0 to 84. The higher the score, the more severe the pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, PhD, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to leigh.charvet@nyulangone.org To gain access, data requestors will need to sign a data access agreement.